CLINICAL TRIAL: NCT03010592
Title: Studying the Airway Microenvironment in Patients Undergoing Surgical and Bronchoscopic Interventions for COPD
Acronym: COPD-ENVIRON
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 217587
Record Dates: First submitted 2016-12-20; First posted 2017-01-05 (Estimated); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Chronic Obstructive Pulmonary Disease; Emphysema; Chronic Bronchitis
Keywords: Lung volume reduction treatment; Endobronchial cryotherapy; Microvesicles
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Bronchitis, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Studying the airway microenvironment in patients undergoing surgical and bronchoscopic interventions for COPD

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is an umbrella term encompassing two entities causing progressive and ultimately disabling breathlessness. Emphysema is a process destructive of the airspaces distal to the terminal bronchioles, with loss of gas exchange tissue, of elastic recoil and of circumferential tethering of the small airways leading to their collapse on forced expiration. Chronic bronchitis is a disorder of the bronchi causing excess production and impaired mobilisation of mucus. Increased parasympathetic tone and progressive remodelling of airways impairs response to bronchodilators. Static and dynamic hyperinflation ensue - a persistently expanded chest and flattened diaphragms despite increasing use of accessory respiratory muscles - resulting in a disadvantaged respiratory pump.

Patients with severe emphysema and hyperinflation benefit from lung volume reduction techniques designed to reduce gas trapping and to improve airflow, chest wall and lung mechanics. The best evidence exists for lung volume reduction surgery (LVRS), which however is not without risk and there is increasing interest in the development of bronchoscopic lung volume reduction (BLVR) techniques including emplacement of endobronchial valves and coils and targeted lung denervation (TLD), which have all been shown to improve lung function, exercise capacity, and quality of life.

Endobronchial cryotherapy is a novel investigational treatment in patients with chronic bronchitis. Porcine models have shown ablation of abnormal metaplastic goblet cells and regeneration of healthy ciliated epithelium and submucosa within 48 hours with complete healing by 60 days following treatment. A pilot study evaluated 11 patients undergoing a lobectomy or pneumonectomy for presumed lung cancer. Metered sprays, one to each of two separate locations, were administered 2 weeks prior to surgery, at least 2cm distal to the proposed resection margin (first segmental and lobular bronchi). No adverse events were reported. Histology of the 8 submitted specimens demonstrated localised cryothermic effect extending to but not beyond the submucosa, and minimal inflammation.

Chronic airway infiltration by neutrophils, macrophages, and Th-1 predominant lymphocytes driven by increased expression of inflammatory proteins, cytokines and chemokines, is intensified during exacerbations. It is generally accepted that acute exacerbations accelerate the decline in lung function in COPD. Recent studies have suggested a role for microvesicles (MVs) in the pathogenesis of COPD, driving exacerbations. MVs are fragments of cell membrane ranging from 0.1 to 1µm in diameter shed by almost all eukaryotic cells. They are recognised to be key mediators of intercellular communication, transporting a variety of molecular cargo including proteins and nucleic acids to distant cells, and have been implicated in various inflammatory diseases including COPD. The majority of studies have looked at circulating endothelial-derived MVs, which are elevated in patients with COPD, are significantly higher during an exacerbation, and are predictive of rapid forced expiratory volume in 1 second (FEV1) decline. However, there is a paucity of data on epithelial-derived MVs within the lung. We know from acute lung injury models that alveolar macrophage-derived microvesicles, which carry biologically active tumour necrosis factor, are rapidly released during the early phase and may play a role in initiating the disease process.

Bronchoalveolar lavage and brushings are established techniques to obtain material for respectively, measurement of inflammatory proteins and microvesicles, and for cytology and messenger ribonucleic acid (mRNA) analysis. A novel technique sampling the mucosal lining fluid using a synthetic absorptive matrix ('bronchosorption') has been shown to have greater sensitivity to standard bronchoalveolar lavage (BAL), eliminating the disadvantage of dilution.

A combination of all three techniques to directly harvest lower airway samples at multiples sites of pulmonary inflammation would allow comparison of proteomic, transcriptomic, and histology data from the endobronchial environment before and after intervention. This would be the first study evaluating the lung microenvironment in this context, which may identify predictive biomarkers of response to intervention and future exacerbation risk.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for lung volume reduction treatment or endobronchial cryotherapy for the management of severe COPD.

Exclusion Criteria:

* Unwilling or unable to sign the informed consent form
* Patients with known Category 3 Organisms as per the Advisory Committee on Dangerous Pathogens (ACDP) for example, Tuberculosis or Human Immunodeficiency Virus.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe COPD who are scheduled to undergo surgical or bronchoscopic lung intervention (n=80)
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2017-02-06 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in airway cytokine levels at 3 months follow-up | Baseline versus 3 months follow-up
  Change in airway cytokine levels measured using a multiplex assay, 3 months following interventional treatment

SECONDARY OUTCOMES:
Association between baseline cytokine levels and future exacerbation frequency at 3 months follow-up | Baseline versus 3 months follow-up
Association between baseline cytokine levels and future decline in lung function at 3 months follow-up | Baseline versus 3 months follow-up
Association between baseline microvesicle levels and future exacerbation frequency at 3 months follow-up | Baseline versus 3 months follow-up
Association between baseline microvesicle levels and future decline in lung function at 3 months follow-up | Baseline versus 3 months follow-up
Change from baseline in airway microvesicle levels at 3 months follow-up | Baseline versus 3 months follow-up
  Change in airway microvesicle levels measured using flow cytometry, 3 months following interventional treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pallav L Shah, MBBS MD FRCP, Principal Investigator — Royal Brompton & Harefields Hospital
Locations (2):
- United Kingdom (2):
  - Chelsea & Westminster Hospital, London, Chelsea
  - Royal Brompton & Harefields Hospital, London, Fulham

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Barnes PJ. Immunology of asthma and chronic obstructive pulmonary disease. Nat Rev Immunol. 2008 Mar;8(3):183-92. doi: 10.1038/nri2254. Epub 2008 Feb 15. PMID 18274560
- [Result] Donaldson GC, Seemungal TA, Bhowmik A, Wedzicha JA. Relationship between exacerbation frequency and lung function decline in chronic obstructive pulmonary disease. Thorax. 2002 Oct;57(10):847-52. doi: 10.1136/thorax.57.10.847. PMID 12324669
- [Result] Takahashi T, Kobayashi S, Fujino N, Suzuki T, Ota C, He M, Yamada M, Suzuki S, Yanai M, Kurosawa S, Yamaya M, Kubo H. Increased circulating endothelial microparticles in COPD patients: a potential biomarker for COPD exacerbation susceptibility. Thorax. 2012 Dec;67(12):1067-74. doi: 10.1136/thoraxjnl-2011-201395. Epub 2012 Jul 27. PMID 22843558
- [Result] Eltom S, Dale N, Raemdonck KR, Stevenson CS, Snelgrove RJ, Sacitharan PK, Recchi C, Wavre-Shapton S, McAuley DF, O'Kane C, Belvisi MG, Birrell MA. Respiratory infections cause the release of extracellular vesicles: implications in exacerbation of asthma/COPD. PLoS One. 2014 Jun 27;9(6):e101087. doi: 10.1371/journal.pone.0101087. eCollection 2014. PMID 24972036
- [Result] Raposo G, Stoorvogel W. Extracellular vesicles: exosomes, microvesicles, and friends. J Cell Biol. 2013 Feb 18;200(4):373-83. doi: 10.1083/jcb.201211138. PMID 23420871
- [Result] Nieri D, Neri T, Petrini S, Vagaggini B, Paggiaro P, Celi A. Cell-derived microparticles and the lung. Eur Respir Rev. 2016 Sep;25(141):266-77. doi: 10.1183/16000617.0009-2016. PMID 27581826
- [Result] Gordon C, Gudi K, Krause A, Sackrowitz R, Harvey BG, Strulovici-Barel Y, Mezey JG, Crystal RG. Circulating endothelial microparticles as a measure of early lung destruction in cigarette smokers. Am J Respir Crit Care Med. 2011 Jul 15;184(2):224-32. doi: 10.1164/rccm.201012-2061OC. Epub 2011 Mar 11. PMID 21471087
- [Result] Thomashow MA, Shimbo D, Parikh MA, Hoffman EA, Vogel-Claussen J, Hueper K, Fu J, Liu CY, Bluemke DA, Ventetuolo CE, Doyle MF, Barr RG. Endothelial microparticles in mild chronic obstructive pulmonary disease and emphysema. The Multi-Ethnic Study of Atherosclerosis Chronic Obstructive Pulmonary Disease study. Am J Respir Crit Care Med. 2013 Jul 1;188(1):60-8. doi: 10.1164/rccm.201209-1697OC. PMID 23600492
- [Result] Takahashi T, Kobayashi S, Fujino N, Suzuki T, Ota C, Tando Y, Yamada M, Yanai M, Yamaya M, Kurosawa S, Yamauchi M, Kubo H. Annual FEV1 changes and numbers of circulating endothelial microparticles in patients with COPD: a prospective study. BMJ Open. 2014 Mar 6;4(3):e004571. doi: 10.1136/bmjopen-2013-004571. PMID 24604485
- [Result] Soni S, Wilson MR, O'Dea KP, Yoshida M, Katbeh U, Woods SJ, Takata M. Alveolar macrophage-derived microvesicles mediate acute lung injury. Thorax. 2016 Nov;71(11):1020-1029. doi: 10.1136/thoraxjnl-2015-208032. Epub 2016 Jun 10. PMID 27287089
- [Result] Leaker BR, Nicholson GC, Ali FY, Daudi N, O'Connor BJ, Barnes PJ. Bronchoabsorption; a novel bronchoscopic technique to improve biomarker sampling of the airway. Respir Res. 2015 Sep 4;16(1):102. doi: 10.1186/s12931-015-0268-5. PMID 26338015